CLINICAL TRIAL: NCT05303012
Title: International, Prospective Multicentre Study to Record the Mental and Physical Effects of the COVID-19 Pandemic on Two Obese Patient Cohorts Pre- and Post-bariatric Surgery (COBESITY-Study)
Brief Title: Multicentre Study to Record the Mental and Physical Effects of the COVID-19 Pandemic (COBESITY-Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-100673
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic; Overweight and Obesity
MeSH Terms: conditions — COVID-19; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight and obese patient cohort: * Age: 18 years and older
  * BMI ≥ 25kg/m²
- Overweight and obese patient cohort with bariatric surgery: * Age: 18 years and older
  * BMI ≥ 25kg/m²
  * Status post sleeve or gastric bypass surgery

SUMMARY:
Prospective, international multicenter study to investigate the physical and psychological effects of the COVID-19 pandemic in two obese patient cohorts (BMI ≥ 25 kg/m²) pre- and post-bariatric surgery. In addition, the investigation of country-specific differences will be performed.

DETAILED DESCRIPTION:
The COVID-19 pandemic, first reported in November 2019, has led to a global health systems emergency. The number of confirmed COVID-19-associated deaths, according to WHO, is higher in countries with high obesity prevalence. However, whether obesity is an independent risk factor of the severity of COVID-19 remains unclear.

Obesity represents one of the major health problems worldwide and the COVID-19 pandemic is expected to further increase obesity prevalence rates. Initial research indicates that the pandemic has also led to an increased incidence and/or worsening of depression and eating disorders. Additional weight gain due to the COVID-19 pandemic may be suspected to increase the prevalence of psychological comorbidities in patients before weight-reducing surgery compared to patients who have already undergone weight-reducing surgery.

Therefore, the main aim of this international study is to gain a better understanding of the mental and physical effects of the coronavirus pandemic on obese patients before and after a weight-reducing surgery and use this to develop approaches for solutions. This study also aims to investigate the country-specific differences (Germany vs England) as well as the differences in the mental effects experienced by overweight patients who have or have not been infected with COVID-19.

To achieve these aims, obese patients aged 18 years and older, before and after weight-reducing surgery, will be recruited from the bariatric surgery clinic at King's College Hospital, NHS Trust Foundation as well as from the Medical University Hospital Hamburg-Eppendorf, Germany. Participants will be asked to complete a questionnaire about their health, socio-economic status, and the effects of the COVID-19 pandemic on their physical and mental health. The questionnaire will take 15 minutes to complete and can be done at home or during the patient's appointment at the bariatric surgery clinic to minimise unnecessary travel.

ELIGIBILITY:
Inclusion Criteria:

Overweight and obese patient cohort

* Age: 18 years and older
* BMI ≥ 25kg/m²

Overweight and obese patient cohort with bariatric surgery

* Age: 18 years and older
* BMI ≥ 25kg/m²
* Status post sleeve or gastric bypass surgery

Exclusion Criteria:

* Age under 18 years
* Cognitive, mental and/or linguistic limitations to complete the questionnaire independently
* Severe somatic illnesses, such as tumour diseases
* Pregnancy or breastfeeding
* Acute need for treatment due to comorbid mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight and obese patients with or without bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
PHQ-4 | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
  Impact of the COVID-19 pandemic on mental health (measured by PHQ-4, PSS-10, and EDEQ scores) as well as on physical health (measured by Δ BMI (kg/m^2) before and after the onset of the pandemic) in two obese patient cohorts pre- and post- bariatric surgery.
PSS-10 | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
  Impact of the COVID-19 pandemic on mental health (measured by PHQ-4, PSS-10, and EDEQ scores) as well as on physical health (measured by Δ BMI (kg/m^2) before and after the onset of the pandemic) in two obese patient cohorts pre- and post- bariatric surgery.
EDEQ-score | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
  Impact of the COVID-19 pandemic on mental health (measured by PHQ-4, PSS-10, and EDEQ scores) as well as on physical health (measured by Δ BMI (kg/m^2) before and after the onset of the pandemic) in two obese patient cohorts pre- and post- bariatric surgery.
BMI | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
  Impact of the COVID-19 pandemic on mental health (measured by PHQ-4, PSS-10, and EDEQ scores) as well as on physical health (measured by Δ BMI (kg/m^2) before and after the onset of the pandemic) in two obese patient cohorts pre- and post- bariatric surgery.

SECONDARY OUTCOMES:
Country-specific differences of the physical and psychological impact of the COVID-19 pandemic | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
Differences in psychological impact in obese patients pre- and post-bariatric surgery | Before the COVID-19 pandemic vs. since the COVID-19 pandemic
Differences in psychological impact between obese patients with and without COVID-19 infection | Before the COVID-19 pandemic vs. since the COVID-19 pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Pia Roser, MD, Principal Investigator — Medical University Hospital Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No